CLINICAL TRIAL: NCT05231356
Title: Role of Magnetic Resonance Imaging(MRI) in Evaluation of Parkinson's Disease
Brief Title: DTI in Evaluation of Parkinsons Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Alaa, AlaaMohamedAlaa, Assiut University
Other Study IDs: MRI Parkinson disease
Record Dates: First submitted 2022-01-29; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Mri in Parkinsons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2: group 1 with positive signs group 2 with negative signs

SUMMARY:
The aim of this study is to evaluate the role of different magnetic resonance sequences in demonstration of microstructural abnormalities in Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder after Alzheimer disease. PD generally begins with motor symptoms, including bradykinesia , rigidity, resting tremor, and postural instability. PD also includes numerous non-motor symptoms (such as cognitive impairment, depression, sleep behavioral problems, and olfactory dysfunction) (1). The classical neuropathologic hallmark of PD involves the loss of dopaminergic neurons in the substantia nigra (SN), resulting in a decreased dopaminergic output through the cortico-basal ganglia-thalamocortical motor circuit, which causes dysregulation of motor functions (2). Another neuropathologic characteristic of PD is the presence of Lewy bodies (3) and neurites in both neuron bodies and axons, including aggregates of the α-synuclein protein (4). When PD begins, the complex features of motor and non-motor symptoms reflect the progression of underlying pathologies, including α-synuclein immunoreactive inclusions in Lewy bodies; loss of dopaminergic, cholinergic, serotonergic, and noradrenergic projections from the brainstem to the midbrain and basal forebrain; and, finally, to the neocortex (5). Over the course of PD, patients commonly experienced comorbid neuropsychiatric disturbances, including depression, behavioral and cognitive deficits, and dementia, which need to be differentiated from other neurodegenerative causes such as dementia with Lewy bodies (DLB) and Alzheimer's disease. On the other hand, the term "parkinsonism" refers to motor syndromes that also present in PD, including bradykinesia, cogwheel rigidity, resting tremor, a slow shuffling gait, and imbalance. The atypical causes of parkinsonism that mimic idiopathic PD include multiple system atrophy (MSA), progressive supranuclear palsy (PSP), or corticobasal syndrome (CBS), as well as drug-induced parkinsonism and others. In PD, the loss of dopaminergic neurons and the accumulation of Lewy bodies are typically accompanied by damage of neuroglial cells and demyelination of axons with increasing microglia concentration in extracellular spaces. It is therefore plausible that the detection of extracellular microstructural abnormalities in brain regions with dopaminergic neurons and along dopaminergic pathways might be a biomarker of incipient PD(6). As regards our knowledge of PD pathophysiology, recent neuroimaging methods make it possible to investigate anatomy and impact of brain alterations, on the basis of functional, structural and diffusion data acquisitions, three complementary techniques to assess brain changes related to neurodegenerative diseases like PD. New MRI techniques and their use in PD and explains how these techniques may be used to detect changes in the brain of PD patients and their relationships with Parkinsonian symptoms. Brain MRI is commonly used in clinical practice to evaluate structural brain anatomy and pathology. In neurodegenerative pathology, brain MRI can identify patterns of structural degradation in order to help make the correct diagnosis. These structural changes can be regions of atrophy or structure signal intensity changes. In the diagnostic work-up of patients with parkinsonism, it is recommended to perform brain MRI (13). The main purpose of brain MRI in the work-up of parkinsonism is to assess cerebrovascular damage (vascular parkinsonism), and to exclude other possible but more rare causes of parkinsonism such as multiple sclerosis , normal pressure hydrocephalus or Wilson's disease. Also, it can support the diagnosis of neurodegenerative atypical parkinsonism Resting-state functional Magnetic Resonance Imaging (fMRI) can be used to study brain connectivity and the alterations of functional networks. A recent review of the literature provided interesting insights into the functional alterations in PD (7): mainly, PD induces functional dysfunctions particularly in the sensorimotor, visual and basal ganglia networks. It is reasonable to argue that fMRI data depends on several parameters, such as the dopaminergic medication state (8) or the fMRI acquisition parameters (7). Concerning anatomical MRI, voxel-based morphometry (VBM) can be used to study the volume of gray matter (9). Recent VBM meta-analyses demonstrated a cortical atrophy in PD patients in the left inferior frontal gyrus, superior temporal gyrus, insula and parietal areas (for a review, see (10)(11) (12), but also in the left-sided parahippocampal gyrus, insula and superior temporal gyrus in younger patients, as well as a correlation between disease duration and motor impairment and gray matter reduction in the left inferior frontal gyrus (10). While fMRI allows the study of functional connectivity by assessing neuronal (dys)functioning related to PD, structural MRI adds information regarding anatomical changes, and particularly cortical lesions that are also involved in the disease progression. Functional and structural MRI data contribute to a substantial, but still partial, understanding of PD pathophysiology. In order to enhance this knowledge, DTI allows the study of white fiber integrity, which is also impacted by the neurodegenerative processes

Diffusion Tensor Imaging (DTI), one of the magnetic resonance imaging (MRI) sequences, has been employed to measure white matter microstructural integrity in neurodegenerative diseases, as well as to visualize brain fiber connections via tractography (6). Fractional anisotropy (FA), radial (RD), axial (AD), and mean diffusivity (MD) have been most commonly used to describe the degree of random motion of water molecules on a microscopic scale. Specifically, FA, which measures the directionality of random water motion, has been used to probe nerve fiber arrangements, axonal integrity, and the degree of axonal myelination (13). FA is clinically feasible to deduce the microstructural integrity of brain tissues, especially preferred to oriented tissues, such as white matter and fiber-tract architectures. MD measures the magnitude of water diffusion. A high MD is thought to indicate broad cellular damages including edema and necrosis. MD is used clinically to capture these microstructural alterations in both gray and white matter tissues (14). AD measures the magnitude of diffusion along the main axis, and RD measures the magnitude of transverse diffusion

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients diagnosed clinically with Parkinson's disease (2) No contraindications of MRI

Exclusion Criteria:

* contraindications of MRI (such as claustrophobia or pacemaker installed

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include 50 patients with identified by MRI. A standardized multi-parametric MR protocol will be implemented for all patients. All sequences will be acquired on a 1.5T MR scanner.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Role o Role of magnetic resonance imaging(MRI) in evaluation of Parkinson's disease f magnetic resonance imaging(MRI) in evaluation of Parkinson's disease | baseline
  analysis of the role of MRI and DTI in evaluation of parkinsons disease

CONTACTS AND LOCATIONS:
Overall Officials: ahmed moustafa mohamed, MD, Principal Investigator — Assuit university hospital Radiology department; MOHAMED koreim mahmoud, MD, Principal Investigator — Assuit university hospital Radiology department; SHADY MOHAMED SAFWAT, MD, Principal Investigator — Assuit university hospital psychiatry and neurology department